CLINICAL TRIAL: NCT05686291
Title: Effectiveness of Hybrid Learning Mode of Volunteer Training: A Randomized Controlled Trial
Brief Title: Effectiveness of Hybrid Learning Mode of Volunteer Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Education University of Hong Kong (Other)
Collaborators: Baptist Oi Kwan Social Service (Other)
Responsible Party: Principal Investigator, CHAN Ka Shing Kevin, Associate Professor, Head of Department of Psychology, Education University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2021-2022-0403
Record Dates: First submitted 2023-01-06; First posted 2023-01-17 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Healthy Volunteer
Keywords: Volunteer training; Hybrid learning mode; Mental illness
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Participants in the treatment condition start the online volunteer training immediately after randomization and completed the online module within 2-week. Then they are invited to attend the face-to-face training within 1-week. They will complete the post-intervention assessment right after they finish the face-to-face training, and be invited to participate in an interview.
  Interventions: Behavioral: Hybrid volunteer training programme
- Wait-list control group (No Intervention): Participants in the waitlist control group will wait for 4 weeks without the training and then complete the post-intervention assessment. The waitlist control participants will start training (equivalent to that of the treatment group) immediately after completing the post-intervention assessment.

INTERVENTIONS:
Behavioral: Hybrid volunteer training programme — The volunteer training will consist of a 6-module online course, followed by 5 face-to-face courses, incorporating the key volunteer training components, including Keyes theory, bio-psycho-social model, stress bucket model, recovery model and CHIME model.
  Arms: Treatment group

SUMMARY:
As the effectiveness of the hybrid volunteer training in Hong Kong is under-studied, this experimental study aims to develop a hybrid learning mode of volunteer training that increase volunteering-related self-efficacy and its associated outcomes among volunteer. In particular, this study compares the efficacy of hybrid volunteer training with the wait-list control group.

The volunteer training will consist of a 6-module online course, followed by 5 face-to-face courses. Each module will consist of the key volunteer training component presented in in written or video format. Materials will be presented interactively to facilitate engagement.

DETAILED DESCRIPTION:
Mental illness poses a challenge to public mental health services because of its high prevalence, symptom chronicity, and impacts on patients and society. Although there is a huge amount of need to serve people with mental illness, there is insufficient manpower. There is much empirical evidence to support the volunteer programs for people with mental illness. However, the literature on hybrid volunteer training is mainly focused on teaching and learning in education, and the effectiveness of the hybrid volunteer training in Hong Kong is under-studied. Therefore, The present study aims to compare the efficacy of hybrid volunteer training with the wait-list control group. We hypothesize that (1) participants who receive hybrid volunteer training will increase their self-efficacy of volunteering after the intervention as compared with the wait-list controls; (2) participants from hybrid volunteer training will have better mental health knowledge and less mental health-related stigmatized beliefs and behavior after the intervention as compared with the wait-list controls.

The volunteer training will consist of a 6-module online course, followed by 5 face-to-face courses, incorporating the key volunteer training components, including Keyes theory, bio-psycho-social model, stress bucket model, recovery model and CHIME model. Each module will consist of the key volunteer training component presented in in written or video format. Materials will be presented interactively to facilitate engagement.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong residents
* Age ≥18 years
* Willing to participate in volunteer service
* Being able to read Chinese
* Have a computer, tablet and/or smartphone device with Internet access
* Have a regular email address
* Willing to give informed consent and comply with the trial protocol

Exclusion Criteria:

* Unable to communicate with Cantonese.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Assessment in Self-Efficacy Towards Service on the Self-Efficacy Towards Service (SETS) Scale at Post-intervention Assessment and Follow-up Assessment | Before intervention, Immediately after intervention, and 4 weeks after intervention
  The SETS scale assess the change in a 5-point Likert scale, ranging from strongly disagree (1) to strongly agree (5).
Change from Baseline Assessment in Mental Health-related Knowledge on the Mental Health Knowledge Schedule (MAKS) at Post-intervention Assessment and Follow-up Assessment | Before intervention and Immediately after intervention, and 4 weeks after intervention
  The MAKS assess the change in a 5-point Likert scale, ranging from strongly disagree (1) to strongly agree (5).
Change from Baseline Assessment in Views of Empowerment on the Empowerment Scale at Post-intervention Assessment and Follow-up Assessment | Before intervention and Immediately after intervention, and 4 weeks after intervention
  The Empowerment Scale assess the change in a 9-point scale of agreement, ranging from strongly disagree (1) to strongly agree (9).
Change from Baseline Assessment in View of Recovery on the Recovery Scale at Post-intervention Assessment and Follow-up Assessment | Before intervention and Immediately after intervention, and 4 weeks after intervention
  The Recovery Scale assess the change in a 9-point scale of agreement, ranging from strongly disagree (1) to strongly agree (9).
Change from Baseline Assessment in Mental Health-related Behaviors on the Intended Behaviour subscale of the Reported and Intended Behaviour Scale (RIBS) at Post-intervention Assessment and Follow-up Assessment | Before intervention and Immediately after intervention, and 4 weeks after intervention
  The RIBS assess the change in a 5-point Likert scale, ranging from strongly disagree to engage in the stated behavior (1) to strongly agree with engaging in the stated behavior (5).
Change from Baseline Assessment in Public Attitudes Toward Mental Illness on the Stigma and Acceptance Scale at Post-intervention Assessment and Follow-up Assessment | Before intervention and Immediately after intervention, and 4 weeks after intervention
  The Stigma and Acceptance Scale assess the change in a 6-point Likert scale, ranging from strongly disagree (1) to strongly agree (6).

SECONDARY OUTCOMES:
Change from Baseline Assessment in Psychological Wellbeing on the World Health Organisation-Five Well-Being Index (WHO-5) at Post-intervention Assessment and Follow-up Assessment | Before intervention and Immediately after intervention, and 4 weeks after intervention
  The WHO-5 assess the change in a 6-point Likert scale, ranging from at no time (1) to all of the time (6).
Change from Baseline Assessment in Anxiety Symptom on the General Anxiety Disorder-7 (GAD-7) at Post-intervention Assessment and Follow-up Assessment | Before intervention and Immediately after intervention and 4 weeks after intervention
  The GAD-7 assess the change in a 4-point Likert scale, ranging from not at all (0) to nearly every day (3).
Change from Baseline Assessment in Depressive Symptom on the Patient Health Questionnaire-9 (PHQ-9) at Post-intervention Assessment and Follow-up Assessment | Before intervention and Immediately after intervention, and 4 weeks after intervention
  The PHQ-9 assess the change in a 4-point Likert scale, ranging from not at all (0) to nearly every day (3).
Change from Baseline Assessment in Quality of Life on the Twelve-item short-form (SF-12) health survey at Post-intervention Assessment and Follow-up Assessment | Before intervention and Immediately after intervention, and 4 weeks after intervention
  The SF-12 assesses the change in a combination of 5-point and 3-point Likert scale, ranging respectively from poor/ never (1) to excellent/ very much (5), and never (1) to very much (3).

CONTACTS AND LOCATIONS:
Overall Officials: Kevin, Ka Shing CHAN, Principal Investigator — The Education University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Baptist Oi Kwan Social Service, Hong Kong
  - The Education University of Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No